CLINICAL TRIAL: NCT07245082
Title: Cohort Study of Patients With Type 2 Diabetes
Brief Title: Patients With Type 2 Diabetes
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202507201RINE
Record Dates: First submitted 2025-11-16; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Obesity; Diabetic macular edema; diabetic kidney disease; Diabetic retinopathy; Nutritional status; Physical activity; Peripheral Arterial Occlusive Disease; Body composition; Metabolic Syndrome; Dynapenia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetic Nephropathies; Diabetic Retinopathy; Motor Activity; Peripheral Arterial Occlusive Disease 1; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetes mellitus

DETAILED DESCRIPTION:
This study aims to establish both retrospective and prospective cohorts of patients with type 2 diabetes, enabling long-term follow-up of metabolic factors and related complications (such as cardiovascular disease, nephropathy, and neuropathy), as well as changes in nutritional status and physical function (including dietary habits, body composition, grip strength, and calf circumference). The goal is to identify risk factors that influence clinical outcomes and to provide evidence to support individualized treatment and integrated care strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 or older.
2. Patients diagnosed with type 2 diabetes (based on medical history, diagnostic code, or use of hypoglycemic medication).
3. Participants are willing to participate in the study and have signed the consent form.
4. Participants are able to complete basic assessments (e.g., height, weight, waist circumference, grip strength, calf circumference, body composition, etc.).

Exclusion Criteria:

1. Individuals who cannot understand the study content.
2. Individuals who cannot cooperate with relevant assessments.
3. Other individuals who are clinically deemed unsuitable for participation by the project leader.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will recruit adult participants aged 18 years or older who have been diagnosed with type 2 diabetes mellitus (T2DM), as confirmed by medical history, diagnostic codes, or current use of hypoglycemic medications. Eligible participants must be willing to join the study and provide written informed consent. In addition, they should be able to complete the required baseline assessments, including anthropometric and functional measurements such as height, weight, waist circumference, handgrip strength, calf circumference, and body composition.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2028-08-21 (Estimated); Study Completion 2028-08-21 (Estimated)

PRIMARY OUTCOMES:
Changes in nutritional status and physical function (including dietary habits, body composition, grip strength, and calf circumference) | Everytime after physician's appointment(Usually 3 months).

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Wen Lu, Present Professor, Study Chair — Department of Family Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided